CLINICAL TRIAL: NCT06391398
Title: The Impact of Education Using a Stoma Care Training Belt on Care Skills, Adaptation, Anxiety, and Patient Satisfaction in Patients Undergoing Intestinal Stoma Creation:Randomized Controlled Trial
Brief Title: The Impact of Education Using a Stoma Care Training Belt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hatice ÖNER CENGİZ, Assist. Prof., Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HOCengiz
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Stoma Colostomy; Stoma Ileostomy
Keywords: Ostomy; Education of patients; Anxiety; Patient Satisfaction
MeSH Terms: conditions — Anxiety Disorders; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: parallel-group, randomized controlled trial will be conducted to assess the effect of the Stoma Care Training Belt on patients' stoma care skills, adaptation, anxiety, and satisfaction. A total of 170 patients, with 85 in the intervention group and 85 in the control group, will be included. All patients in the study will receive routine stoma care education as part of their standard treatment and care. In addition to routine treatment and care, patients in the intervention group will receive education with the Stoma Care Training Belt during the preoperative period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stoma care belt group (Experimental): In addition to routine treatment and care, patients in the intervention stoma care belt group will receive education with the Stoma Care Training Belt during the preoperative period.
  Interventions: Behavioral: Stoma care education with the Stoma Care Training Belt
- Control group (No Intervention): Patients in the control group will not undergo any additional intervention beyond routine treatment and care.

INTERVENTIONS:
Behavioral: Stoma care education with the Stoma Care Training Belt — Stoma care education
  Arms: Stoma care belt group

SUMMARY:
Intestinal stoma is a surgical procedure performed to create an artificial opening in the intestine. To improve the quality of life of individuals with stoma, it is essential to address physiological and psychosocial issues and ensure adaptation to the stoma. Patient education on stoma care during the preoperative period may facilitate stoma adaptation. The aim of this study is to evaluate the impact of the education provided to patients undergoing intestinal stoma creation using a Stoma Care Training Belt on stoma care skills, adaptation, anxiety, and satisfaction.

DETAILED DESCRIPTION:
Introduction:Intestinal stoma is a surgical procedure performed to create an artificial opening in the intestine. To improve the quality of life of individuals with stoma, it is essential to address physiological and psychosocial issues and ensure adaptation to the stoma. Patient education on stoma care during the preoperative period may facilitate stoma adaptation. The aim of this study is to evaluate the impact of the education provided to patients undergoing intestinal stoma creation using a Stoma Care Training Belt on stoma care skills, adaptation, anxiety, and satisfaction. This study will be conducted as a parallel group, randomized controlled study at Ankara University Health Practice and Research Hospitals Ibn-i Sina Research and Practice Hospital and Ankara University Health Practice and Research Hospitals Cebeci Research and Practice Hospital General Surgery Clinics.The analysis was performed in G*Power version 3.1.9.4.It was planned to include a total of 170 patients in the study, 85 patients in each group.In order to ensure similarity between groups; Simple randomization will be used to assign the women in the sample group to the experimental and control groups. Data, sociodemographic and medical data form, State Anxiety Scale, Stoma Care Skill Rubric, Ostomy Adaptation Scale-23 and Visual Analogue Scale (VAS)-Patient satisfaction level will be collected.Patients will be evaluated 5 times in total: on the day of discharge, and on the 5th, 15th and 30th days after discharge. The data will be evaluated in a computer environment with appropriate statistical methods using the Statistical Package for Social Sciences 25 (SPSS) for Windows statistical package program.Ethics committee permission was received for the research from Ankara University Ethics Committee. Permission was obtained from the institution where the research would be conducted.This research is supported by the Scientific and Technological Research Council of Turkey (TUBITAK).

ELIGIBILITY:
Inclusion Criteria:

* Intestinal stoma (colostomy or ileostomy) opened for the first time,
* Those aged 18 and over, Able to speak and understand Turkish,
* Conscious, oriented and cooperative,
* Does not have a diagnosed psychiatric or psychological disease,
* There is no obstacle to stoma care, Those who have no previous stoma knowledge or training.

Exclusion Criteria:

* Those who do not agree to participate in the study,
* Refuses to perform stoma care in the postoperative period,
* Leaving the job voluntarily, Those who died during the work process,
* Referred from the relevant hospital during the treatment process,
* Any postoperative complications (bleeding, infection, fistula, etc.) develop,
* Data collection forms could not be completed,
* Patients who cannot be reached will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Stoma Care Skills | day of discharge and on days 5th, 15th and 30th after discharge
  Stoma Care Skill will be evaluated 4 times in total, using the Stoma Care Skill Rubric, on the day of discharge, and on the 5th, 15th and 30th days after discharge. On the relevant days, patients come to the polyclinic for control. It consists of 23 items that include stoma care process steps. For each process step, the learner's competence is scored between 0-2 (0- Insufficient, 1- Partially adequate, 2- Satisfactory). A minimum of 0 and a maximum of 46 points can be obtained from the key. The total score obtained from the key indicates the adequacy of stoma care skills.
Stoma compliance | day of discharge and on days 5th, 15th and 30th after discharge
  Patients' stoma compliance levels will be evaluated 4 times in total, using the Ostomy Compliance Scale-23, on the day of discharge and on the 5th, 15th and 30th days after discharge. On the relevant days, patients come to the polyclinic for control. The total score obtained from the scale varies between 20-80. A high score indicates a high level of anxiety, and a small score indicates a low level of anxiety. The scale score varies between 0-92 points. Higher scores from each scale item indicate increased compliance.
Anxiety | the day before surgery, day of discharge and on days 5th, 15th and 30th after discharge
  The anxiety levels of the patients will be evaluated 5 times in total, using the State Anxiety Scale, on the day before surgery, on the day of discharge, and on the 5th, 15th and 30th days after discharge. On the relevant days, patients come to the polyclinic for control.The total score obtained from the scale varies between 20-80. A high score indicates a high level of anxiety, and a small score indicates a low level of anxiety.

SECONDARY OUTCOMES:
Patient Satisfaction | the day before surgery, day of discharge
  Visual Analog Scale will be used to evaluate patients' satisfaction levels with the training provided with the Stoma Care Training Belt. Accordingly, they will be asked to give a score between 0 (very dissatisfied) and 10 (highest possible satisfaction) regarding their level of satisfaction with the training provided with the Stoma Care Training Belt. As the score increases, the satisfaction level increases.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet YÜKSEKKAYA, PhD, Study Chair — Ankara University; İlknur Münevver GÖNENÇ, PhD, Study Chair — Ankara University; Ayten DEMİR, PhD, Study Chair — Ankara University; Ayhan Bülent ERKEK, MD, Study Chair — Ankara University; Şiyar ERSÖZ, MD, Study Chair — Ankara University; Serpil UÇAR, MSc, Study Chair — Ankara University
Locations (2):
- Turkey (Türkiye) (2):
  - Hatice ÖNER CENGİZ, Altındağ, Ankara
  - Ankara University, Ankara, Ankara

IPD SHARING:
Plan to Share IPD: No
The researchers do not intend to share research data. But the researchers may only share data from participants for meta-analysis study of randomized controlled trials.